CLINICAL TRIAL: NCT01445873
Title: NON-INTERVENTIONAL (NI) DRUG STUDY PROTOCOL: THREE-COUNTRY PILOT STUDY FOR RETROSPECTIVE CHART REVIEW OF EFFECTIVENESS OF THELIN® (SITAXSENTAN) IN PATIENTS WITH PULMONARY ARTERIAL HYPERTENSION (PAH)
Brief Title: Pilot Chart Review Study Of Sitaxentan Sodium (Thelin) In Patients With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1321051
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; sitaxentan sodium; Thelin
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAH patients receiving Sitaxentan
  Interventions: Drug: Sitaxentan sodium

INTERVENTIONS:
Drug: Sitaxentan sodium — Sitaxentan sodium 100 mg / day

SUMMARY:
The objectives of this study are to develop research methods and corresponding materials for a study of the effectiveness of sitaxentan sodium (Thelin) in "real-world" settings; to pilot test these methods at three study centers in Europe; and to refine and finalize research methods and corresponding materials for possible use in a follow-on, full-scale examination of the effectiveness of sitaxentan sodium (Thelin) in "real-world" settings.

DETAILED DESCRIPTION:
At each centre, approximately 12-15 Pulmonary Arterial Hypertension (PAH) consecutive patients who have received Thelin and who meet all other study entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PAH, or PAH secondary to connective tissue disease
* Receipt of Thelin for treatment of PAH
* 6 months of follow-up (except in the event of death) subsequent to initial receipt of Thelin
* Minimum of one clinic visit documented in the medical record during the 6-month period subsequent to initial receipt of Thelin

Exclusion Criteria:

* Participation in any investigational study of Thelin or any other medication for the treatment of PAH during the period beginning 6 months prior to initial receipt of Thelin and ending 6 months subsequent to such receipt
* Receipt of Thelin prior to January 11, 2005 (i.e., the date following the last day on which patients could be enrolled in double-blind treatment in STRIDE-1, STRIDE-2, and/or STRIDE-6); or
* Known contraindications to Thelin therapy (i.e., known hypersensitivity to sitaxsentan or any of its excipients; mild-to-severe hepatic impairment [Child-Pugh Class A-C]; elevated aminotransferases prior to initiation of treatment, defined as aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] >3 times upper limit of normal [ULN]; concomitant use of cyclosporin A; lactation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Pulmonary Arterial Hypertension (PAH) (Idiopathic or secondary to connective tissue disease), receiving sitaxentan sodium (Thelin) for treatment of their PAH for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2011-03-28 (Actual); Study Completion 2011-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321051&StudyName=Pilot%20Chart%20Review%20Study%20Of%20Sitaxentan%20Sodium%20%28Thelin%29%20In%20Patients%20With%20Pulmonary%20Arterial%20Hypertension%20%28PAH%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data for this retrospective non-interventional study were abtracted from the medical records of subjects who met study entry criteria.
Pre-assignment Details: Patterns of treatment with Thelin including duration and daily dosages reflect treament participants received in clinical practice. Treatment was not specified by the protocol.
Groups:
- Sitaxentan (Thelin): Duration and dose as prescribed in clinical practice.
Period: Overall Study
Arm/Group | Sitaxentan (Thelin)
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
Age, Customized [Count of Participants; unit: Participants]
  19 to 24 years | 0
  25 to 30 years | 2
  31 to 36 years | 2
  37 to 42 years | 1
  43 to 48 years | 2
  49 to 54 years | 4
  55 to 60 years | 2
  61 to 66 years | 5
  67 to 72 years | 9
  73 to 78 years | 7
  79 to 84 years | 1
  85 to 90 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Patterns of Pharmacotherapy With Sitaxentan Sodium (Thelin): Mean Time to Therapy Augmentation
Description: Participants still receiving Thelin with evidence of receipt of another PAH-related therapy (eg. bosentan, sildenafil) not previously received during the study period. Mean time in months to therapy augmentation.
Time Frame: Day 1 to Month 6
Population: Full analysis set (FAS): participants with idiopathic pulmonary arterial hypertension (PAH) or PAH secondary to connective tissue disease, receipt of Thelin for treatment of PAH, 6 months of follow-up (except for death) after initial receipt (IR) of Thelin, and at least 1 clinic visit in medical record during 6-month period after IR of Thelin.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
months | 2.2 (1.2)

2. Primary Outcome: Patterns of Pharmacotherapy With Sitaxentan Sodium (Thelin): Therapy Switching
Description: Participants with evidence of discontinuation of Thelin therapy and evidence of receipt of another PAH-related therapy not previously received during the study period.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
participants | 0

3. Primary Outcome: Patterns of Pharmacotherapy With Sitaxentan Sodium (Thelin): Therapy Discontinuation
Description: Participants were designated as having discontinued Thelin therapy if there was evidence in the medical records that treatment had been terminated.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
participants | 0

4. Primary Outcome: Patterns of Pharmacotherapy With Sitaxentan Sodium (Thelin): Therapy Duration
Description: Duration of Thelin therapy based on time from index date (Day 1 of treatment) until the date of discontinuation of Thelin therapy.
Time Frame: Day 1 to Month 6
Population: FAS; participants without evidence of discontinuation of Thelin therapy were censored at the end of follow-up (at 6 months or death if prior to 6 months).
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
months | 6 (0)

5. Primary Outcome: Patterns of Pharmacotherapy With Sitaxentan Sodium (Thelin): Numbers of Therapy-days Dispensed
Description: Duration of Thelin therapy from initial receipt until date of discontinuation of thelin therapy or the end of follow-up, whichever occurred first.
Time Frame: Day 1 to Month 6
Population: Not analyzed: duration of Thelin therapy as number of therapy days dispensed was not summarized; this measure was reported as duration in months only.
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 0

6. Primary Outcome: Patterns of Pharmacotherapy With Sitaxentan Sodium (Thelin): Daily Dosage
Description: Daily dosage of Thelin based on information in the medical record for the baseline visit and all follow-up clinic visits.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
mg | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Use of Other Pulmonary Arterial Hypertension (PAH)-Related Medications
Description: Use of PAH-related medications other than Thelin described by class of agent received.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
percentage of participants
  Anticoagulants | 83.3
  Diuretics | 88.9
  Calcium channel blockers | 22.2
  Digoxin | 5.6
  Supplemental oxygen | 44.4
  Prostanoids | 27.8
  Other endothelin receptor antagonists | 0.0
  Phosphodiesterase-5 inhibitors | 47.2

8. Secondary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class of Pulmonary Hypertension
Description: Class I: no limitation of usual (usl) physical activity (PA); PA does not increase(d) (incr) dyspnea (dys), fatigue (ftg), chest pain (CP), or syncope (syn); Class II: mild limitation of usl PA; no discomfort at rest, but normal PA causes incr dys, ftg, CP, or presyncope (presyn); Class III: marked limitation of PA; no discomfort at rest but < ordinary activity causes incr dys, ftg, CP, or presyn; Class IV: unable to perform any PA at rest; may have signs of right ventricular failure; sys and/or ftg at rest and symptoms are incr by almost any PA.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index (prior to Thelin initiation) and ≥ 1 WHO value recorded during follow-up.
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 32
participants
  Pre-index functional class (FC) I to FC I | 0
  Pre-index functional class (FC) I to FC II | 0
  Pre-index functional class (FC) I to FC III | 0
  Pre-index functional class (FC) I to FC IV | 0
  Pre-index functional class (FC) II to FC I | 0
  Pre-index functional class (FC) II to FC II | 1
  Pre-index functional class (FC) II to FC III | 2
  Pre-index functional class (FC) II to FC IV | 0
  Pre-index functional class (FC) III to FC I | 0
  Pre-index functional class (FC) III to FC II | 4
  Pre-index functional class (FC) III to FC III | 17
  Pre-index functional class (FC) III to FC IV | 3
  Pre-index functional class (FC) IV to FC I | 0
  Pre-index functional class (FC) IV to FC II | 0
  Pre-index functional class (FC) IV to FC III | 3
  Pre-index functional class (FC) IV to FC IV | 2

9. Secondary Outcome: Change From Baseline in Mean Right Atrial Pressure
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and ≥ 1 value recorded during follow-up period.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 3
mm Hg | -1.3 [-3.9 to 1.2]

10. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: Data not analyzed: no participants had pre-index and follow-up values reported for this outcome measure.
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and follow-up values.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 3
mm Hg | 3.0 [0.1 to 5.9]

12. Secondary Outcome: Change From Baseline in Left Ventricular End Diastolic Pressure
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: Data not analyzed: no participants had pre-index and follow-up values for this outcome measure.
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and follow-up value.
Measure: Mean (95% Confidence Interval); unit: Dyn/s/cm5
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 3
Dyn/s/cm5 | -214.3 [-419.1 to -9.6]

14. Secondary Outcome: Change From Baseline in Cardiac Output
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and follow-up value.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 2
L/min | 0.4 [-1.2 to 1.9]

15. Secondary Outcome: Change From Baseline in Tei Index
Description: Difference between pre-index and follow-up value. Combined myocardial performance index calculated by adding isovolumic contraction time and isovolumic relaxation time and dividing the resulting sum by ejection time.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and ≥ 1 follow-up value.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 8
ratio | -0.1 [-0.3 to 0.0]

16. Secondary Outcome: Change From Baseline in Tricuspid Regurgitant Velocity
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and ≥ 1 follow-up value.
Measure: Mean (95% Confidence Interval); unit: m/sec
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 19
m/sec | -0.3 [-0.5 to 0.0]

17. Secondary Outcome: Change From Baseline in the Total Distance Walked During 6 Minute Walk Test (6MWT)
Description: 6MWT was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety. Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with pre-index and 1 value recorded during follow-up period.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 30
meters | 28.5 [4.7 to 52.3]

18. Secondary Outcome: Change From Baseline in Borg Dyspnoea Score
Description: Borg dyspnoea scale is a 10-point scale where following scores stands for severity of dyspnoea: 0 (no breathlessness at all); 0.5 (very very slight [just noticeable]); 1 (very slight); 2 (slight breathlessness); 3 (moderate); 4 (some what severe); 5 (severe breathlessness); 7 (very severe breathlessness); 9 (very very severe [almost maximum] and 10 (maximum). Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with ≥ 1 value recorded during follow-up period.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 27
units on a scale | 4.9 [4.0 to 5.7]

19. Secondary Outcome: Change From Baseline in Percent of Predicted Peak VO2
Description: Difference between pre-index and follow-up value.
Time Frame: Baseline to Month 6
Population: FAS; N=number of participants with ≥ 1 value recorded during follow-up period.
Measure: Mean (95% Confidence Interval); unit: percent Vo2
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 2
percent Vo2 | 3.5 [0.3 to 6.7]

20. Secondary Outcome: Pulmonary Arterial Hypertension (PAH) Severity and Functional Status: Time to Clinical Worsening
Description: Occurrence of any of the following: death, unplanned PAH-related hospitalization, initiation of epoprostenol, arterial septostomy, lung or heart/lung transplantation, ≥15% decrease from baseline in 6 minute walk test, signs/symptoms of right sided heart failure, and/or worsening WHO functional class.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
months | 2.8 (1.6)

21. Secondary Outcome: Other Pulmonary Arterial Hypertension (PAH)-Related Outcomes: Mortality
Description: Number of participants who died during the follow-up period.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
participants | 0

22. Secondary Outcome: Number of Hospitalizations
Description: All hospitalizations during the follow-up period recorded in medical records.
Time Frame: Day 1 to Month 6
Population: FAS
Measure: Mean (95% Confidence Interval); unit: hospitalizations
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 36
hospitalizations | 0.5 [0.3 to 0.8]

23. Secondary Outcome: Other Pulmonary Arterial Hypertension (PAH)-Related Outcomes: Lung Transplantation
Description: Number of participants who received an lung transplant during hospitalization.
Time Frame: Day 1 to Month 6
Population: FAS; N=number of participants with hospitalizations during follow-up period.
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 13
participants | 0

24. Secondary Outcome: Other Pulmonary Arterial Hypertension (PAH)-Related Outcomes: Heart/Lung Transplantation
Description: Number of participants who received an heart/lung transplant during hospitalization.
Time Frame: Day 1 to Month 6
Population: FAS; N=number of participants with hospitalizations during follow-up period.
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 13
participants | 0

25. Secondary Outcome: Other Pulmonary Arterial Hypertension (PAH)-Related Outcomes: Atrial Septostomy
Description: Number of participants who received an atrial septostomy (balloon or blade) during hospitalization.
Time Frame: Day 1 to Month 6
Population: FAS; N=number of participants with hospitalizations during follow-up period.
Measure: Number; unit: participants
Arm/Group | Sitaxentan (Thelin)
Number analyzed (Participants) | 13
participants | 0

ADVERSE EVENTS:
Description: Pre-specified AEs of interest reported in medical records. Other events = emergency hospital admission, worsening PAH, unexplained anemia, alopecia, diarrhea, fatigue, obstipation, loss of appetite, gastric pain, numerous defecation, INH out of range, cardial decompensation, joint pain, pre-syncope, infection of IV line with need of explanation.
Arm/Group | Sitaxentan (Thelin)
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 27/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxentan (Thelin) (N=36)
Headache (General disorders) | 3
Peripheral edema (General disorders) | 15
Nausea (General disorders) | 3
Dizziness (General disorders) | 12
Nasal congestion (General disorders) | 0
Bleeding (General disorders) | 5
Other events (General disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.